CLINICAL TRIAL: NCT02334618
Title: Clinical Trial of an Insole Sensor to Determine Optimal Limb Loading in the Rehabilitation of Ankle Fractures
Brief Title: Insole Sensor to Determine Optimal Limb Loading in the Rehabilitation of Ankle Fractures
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Rothberg, M.D., University of Utah
Other Study IDs: 73982
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-08

CONDITIONS: Ankle Fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to use a novel load monitoring technology to correlate limb loading to ankle fracture outcomes. This study will collect continuous limb loading data and will provide the first objective insight into how limb loading directs fracture healing.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has an ankle fracture
* Patient speaks English
* Patient weighs between 100 and 250 pounds
* Patient lives in close enough proximity to the hospital to return for all appointments (~100 miles)

Exclusion Criteria:

* Patient is younger than 18 years of age
* Patient has multiple fractures that would alter weight bearing protocol
* Patient does not speak English
* Patient weighs less than 100 pounds or more than 250 pounds
* Patient does not live in close enough proximity to the hospital to return for all appointments (~>100 miles)
* Patient has a traumatic brain injury that would make it so they cannot consent
* Patient has diabetes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the University of Utah emergency department with ankle fractures.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-08; Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Patient Activity Measure (PAM-13) Questionnaire | Follow Up Visits up to 1-Year
  A subjective evaluation of perceived compliance with physician instructions

SECONDARY OUTCOMES:
X-ray (AP and Lateral) | Follow Up Visits up to 1-Year
  Subjectively evaluate fracture healing

CONTACTS AND LOCATIONS:
Overall Officials: David Rothberg, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopedics Center, Salt Lake City, Utah, United States